CLINICAL TRIAL: NCT01568736
Title: B7 Coreceptor Molecules as Clinically-Relevant Surrogate Biomarkers in the Hyper IgD Syndrome (HIDS) Form of Mevalonate Kinase Deficiency (MKD)
Brief Title: B7 Coreceptor Molecules in Hyper IgD Syndrome Form of Mevalonate Kinase Deficiency
Acronym: HIDS-MKD
Status: Withdrawn | Type: Observational
Why Stopped: never started
Sponsor: Michigan Technological University (Other)
Responsible Party: Sponsor
Other Study IDs: STAIR 7003
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2012-03

CONDITIONS: Hyper IgD Syndrome; Mevalonate Kinase Deficiency
Keywords: Hyper IgD Syndrome (HIDS); Mevalonate Kinase Deficiency (MKD)
MeSH Terms: conditions — Mevalonate Kinase Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The hyper IgD syndrome (HIDS) is an inflammatory disease caused by mevalonate kinase deficiency. There is no cure, and available treatments of HIDS febrile episodes have shown limited clinical efficacy. The development of effective interventions for HIDS is limited by our poor understanding of the disease. The goal of the study is to better characterize the inflammatory response during HIDS episodes and to determine the relationship between this response and blood and urine markers of mevalonate kinase deficiency. This knowledge will help us learn more about the cause of the disease and should lead to the identification of new disease biomarkers that can be used to evaluate clinical efficacy in future therapeutic trials.

The primary hypothesis is that the costimulatory B7 glycoprotein abnormalities identified in the murine MKD model will be recapitulated in sera obtained from human HIDS patients, either before, during or after febrile episodes. The secondary hypothesis is that B7 glycoprotein molecule levels will correlate with clinical symptomatic severity score, other known biomarkers of HIDS, markers of inflammation and or markers of isoprenoid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* any race or ethnicity
* diagnosed with HIDS

Exclusion Criteria:

* parents' inability to donate blood
* currently having cancer, renal failure, diabetes, liver disease, thyroid diseases, major infectious diseases or immunodeficiency
* pregnancy
* inability to provide consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Hyper IgD Syndrome (HIDS)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Michigan Techinical University, Houghton, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Oregon Health & Science University, Portland, Oregon
- Radbound University of Nijmegen Medical Centre, Nijmegen, Netherlands